CLINICAL TRIAL: NCT01171157
Title: An Observational Case Control Study of Effectiveness of Influenza Vaccination and Burden of Illness in Community-dwelling Elderly With Influenza-like Illness in Southern Brazil
Brief Title: Effectiveness of Flu Vaccination and Burden of Illness Among Community-dwelling Elderly With Influenza Like Illness in Brazil
Status: Terminated | Type: Observational
Why Stopped: In the context of the World Health Organization's (WHO) Phase 6 pandemic influenza declaration the conduct of the study was deemed no longer feasible
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112868
Record Dates: First submitted 2010-07-15; First posted 2010-07-28 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: Influenza-like illness; vaccine effectiveness; elderly; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One nose/throat swab

GROUPS / COHORTS (1):
- Group 1: Subjects with influenza like illness
  Interventions: Other: Routine sample collection

INTERVENTIONS:
Other: Routine sample collection — Collection of routine nasal/throat swab samples

SUMMARY:
The purpose of this research study is to estimate how many elderly people who have symptoms that look like influenza (i.e. an influenza-like illness) actually have the disease and how effective influenza vaccines are in preventing influenza in elderly people. The study will also examine the severity of the disease (e.g. how long are people ill, were there any complications) and how it affects everyday life (e.g. cost, medications, care by family members).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female >= 65 years of age.
* Written informed consent obtained from the subject.
* Presenting within the first 72 hours of an influenza-like illness. Influenza-like illness is defined as the presence of:

  * Fever measured by the patient or physician and at least one of the following symptoms:
  * Sore throat.
  * Coryza (runny nose) and/or nasal congestion.
  * Cough.
* Availability to be followed up by phone or in person after an interval of approximately 14 - 21 days.

Exclusion Criteria:

* Receipt of any experimental influenza vaccine within 6 months of the onset of the influenza-like illness.
* Terminal stage of disease.
* Subjects living in a nursing home.
* Use of any investigational or non-registered product planned during the study period.
* Subjects who have already been enrolled in this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged 65 years and over, consulting a physician for an influenza-like illness during the influenza season.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-05-26; Primary Completion 2009-06-01 (Actual); Study Completion 2009-06-29 (Actual)

PRIMARY OUTCOMES:
Laboratory-confirmed influenza status in patients presenting with influenza-like illness defined as positive for PCR for influenza A or B | At enrolment (day 0)

SECONDARY OUTCOMES:
Number of days of illness since onset of influenza-like illness | At the follow-up contact (between day 12 and 28)
Number of days of reduced activity since onset of influenza-like illness | At the follow-up contact (between day 12 and 28)
Number of days off work of other family members or caregivers to provide patient care since onset of influenza-like illness | At the follow-up contact (between day 12 and 28)
Number of medical visits related to influenza-like illness since Visit 1 | At the follow-up contact (between day 12 and 28)
Use of medication since onset of influenza-like illness | At the follow-up contact (between day 12 and 28)
Occurrence of complications since onset of influenza-like illness | At the follow-up contact (between day 12 and 28)
Hospitalization since onset of influenza-like illness | At the follow-up contact (between day 12 and 28)
Presence of non-influenza respiratory pathogens in patients presenting with influenza-like illness defined as positivity by PCR | At enrolment (day 0)
Number of deaths | At the follow-up contact (between day 12 and 28)
Clinical features related to influenza-like illness | At enrolment (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Curitiba/Paraná, Paraná, Brazil